CLINICAL TRIAL: NCT06257329
Title: Epidemiological, Clinical and Biological Characteristics and Therapeutic Management of ICU Patients With Severe Acute Exacerbation of COPD. Evaluation of Prognosis and Factors Associated With Survival.
Brief Title: Patients With Severe Acute Exacerbation of COPD Ans Admitted in ICU Register.
Acronym: COPDregister
Status: Recruiting | Type: Observational
Sponsor: Alexis FERRE (Other)
Responsible Party: Sponsor-Investigator, Alexis FERRE, coordinating investigator, Versailles Hospital
Organization: Versailles Hospital (Other)
Other Study IDs: P22/13_BPCO register
Record Dates: First submitted 2024-02-06; First posted 2024-02-13 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: COPD Exacerbation
MeSH Terms: interventions — Registries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: register — Multicentre prospective observational register

SUMMARY:
The objective of this prospective observational study is to describe the epidemiological, clinical and biological characteristics of admitted patients in ICU for severe acute exacerbation of COPD, to assess the different therapeutics used, to evaluate the prognosis of patients with short, medium and long term ( 1 year) and the various factors associated with survival in ICU

DETAILED DESCRIPTION:
This is a prospective study for which data will be collected from pseudonymised. General information on the research activity clinic of the Intensive Care Service of the CH of Versailles is provided by poster, patient booklet or debrief hospitalization, indicating to relatives and/ or patients their possible participation in retrospective or prospective studies.

This research is conducted in accordance with the reference methodology MR 004 approved by the National Commission of Informatics and Libertés (CNIL) and to which the Centre hospitalier de Versailles is committed to comply. For this purpose, an information note will be given to each patient participating in this project in order to seek its non-opposition of participation in this study.

This prospective study is based solely on the examination of files medical. The data collected are only non-sensitive medical data.

This study complies with legal and regulatory requirements. In addition, this research project was submitted to the Ethics Committee (EC) of the Société de Réanimation de Langue Française (SRLF) who gave an opinion favorable on 06/10/2022 (Registration number referenced: CE SRLF 22- 056).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 40 years old
2. COPD documented or strongly suspected

   * Chronic respiratory symptoms (dyspnoea, cough and/or sputum)
   * Exposure to a known risk factor for COPD (such as tobacco smoke)
   * If available, respiratory function tests showing non- or partially reversible obstructive syndrom (post-bronchodilator ratio FEV1/CV < 0.7)
3. Severe acute exacerbation, defined as a worsening of the patient's usual respiratory symptoms with signs of acute respiratory distress (polypnoea ≥ 30 cycles.min-1 or use of accessory respiratory muscles) and/or hypercapnic acidosis (with PaCO2 ≥ 45 mmHg and pH ≤ 7.35)
4. Admission to an ICU, a step-up unit or a respiratory care unit

Exclusion Criteria:

1. Known asthma (according to the criteria of the international "Global initiative for asthma" guidelines)
2. Patient refusal to participate (information note, application for non-opposition)

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with severe acute exacerbation of COPD admitted in ICU
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2027-10-01 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
the epidemiological, clinical and biological characteristics of patients admitted to the ICU for a severe acute exacerbation of COPD | 5 year
  to describe the epidemiological, clinical and biological characteristics of patients admitted to the ICU for a severe acute exacerbation of COPD

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Centre hospitalier de Versailles, Le Chesnay
  - CH Le Mans, Le Mans

IPD SHARING:
Plan to Share IPD: Undecided